CLINICAL TRIAL: NCT01148628
Title: Dose-finding Study of CAELYXTM and RAD001 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern Europe New Drug Organization (Other)
Collaborators: Novartis (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S065RDCX01
Record Dates: First submitted 2010-06-11; First posted 2010-06-22 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Everolimus; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD 001 in combination with CaelyxTM (Experimental): RAD001 will be given p.o. at increasing doses (no intra-patient)and CaelyxTM will be administered i.v. at a fixed dose.
  At each dose level 3 to 6 patients will be entered, according to toxicities observed; the first 3 patients can be treated simultaneously; subsequent patients can be treated after the first 3 have been observed for at least one cycle (4 weeks).
  The dose escalation process will be discontinued once the MTD has been achieved and the RD will be evaluated in a subsequent expansion part of the study.
  Interventions: Drug: RAD 001 in combination with Caelyx

INTERVENTIONS:
Drug: RAD 001 in combination with Caelyx — RAD001 (tablets; 2.5mg) is administered daily at 5, 7.5, 10 mg. CAELYXTM (vials; 50 mg/25mL)is administered i.v.every 4 weeks at 40mg/m2. One treatment cycle is 4 weeks.

SUMMARY:
This is a dose finding, open-label, uncontrolled, dose-escalation trial to determine the Maximum Tolerated Dose (MTD) and the Recommended Dose (RD) of the combination RAD001 (escalating daily dose) and CaelyxTM (fixed dose) to patients with advanced solid tumors.

Other purposes of the study are:

1. define the safety profile of the combination after repeated administrations
2. define hints of antitumor activity, to be confirmed in subsequent disease-oriented expansion phases at the RD.
3. define the pharmacokinetic profile of the combination

DETAILED DESCRIPTION:
mTOR inhibitors are a new class of targeted antitumor agents which showed interesting antitumor activity in a variety of solid tumors, including prostate, soft tissue sarcomas , ovarian, endometrial, kidney, and breast cancer. They also exert an antiangiogenic effect and are almost devoid of bone marrow toxicity as single agents which makes them suitable for combination with cytotoxic drugs.

Anthracyclines are among the most used and effective cytotoxic agents, and in solid tumors their indications include, among others, breast, ovary, endometrial, prostate cancer. Liposomal Doxorubicin (CaelyxTM) could be an adequate replacement of doxorubicin to avoid potential side effects such as cardiotoxicity, alopecia, GI toxicity.

Testing a combination regimen including mTOR inhibitors and anthracyclines in those tumors which are known to be sensitive to both compounds is of high clinical interest and worthwhile.

ELIGIBILITY:
Inclusion Criteria:

1. Histological/cytological diagnosis of solid tumors types for which treatment with an anthracycline containing combination might be indicated.
2. Documented progressive disease prior to entry in the study
3. Though not a primary endpoint of this study when possible presence of measurable and/or evaluable disease according to modified RECIST criteria (histological/cytological confirmation of the neoplastic nature of a solitary lesion is not required in this dose finding study). For patients with no measurable disease (prostate and ovarian cancer) serum tumor marker (CA125 and PSA) is acceptable.
4. Preferentially ≤ 2 prior chemotherapies for advanced disease
5. An ECOG performance status of 0 or 1
6. Serum cholesterol <350 mg/dL and triglycerides <400 mg/dL
7. Adequate hematological, liver and renal function (hemoglobin ≥ 9g/dL, absolute neutrophil count [ANC] ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L, bilirubin ≤ UNL; alkaline phosphatase ≤ 1.5 x UNL; AST, ALT ≤ UNL or 2.5 x UNL in case of liver metastases; albumin ≥ 2.5 g/dL; creatinine ≤ UNL.
8. Male and female patients who are not surgically sterile or postmenopausal must agree to use reliable methods of birth control for the duration of the study until 30 days after the last dose of study drug
9. Able to understand and give written informed consent
10. Abdomen/Pelvis CT scans in the 4 weeks before planned treatment start
11. HBV/HCV testing in the 2 weeks before treatment start in specific categories of patients with hepatitis B and C risk factors and in additional patients at the discretion of the investigators.

Exclusion Criteria:

1. Prior Caelyx TM
2. Prior anthracycline therapy within last 12 months
3. Patients with endometrial ca. who received both chemotherapy and radiotherapy as palliative treatment. Patients who received both chemotherapy and radiotherapy as adjuvant treatment would be accepted provided that treatment has been completed more than 2 years before inclusion; if treatments has been completed less than 2 years the inclusion will be accepted only after Study Chair's approval.
4. Documented resistance to anthracycline therapy i.e progression whilst on therapy or within 6 months after the end of therapy having achieved a response or stable disease or after adjuvant therapy.
5. Prior cumulative dose of > 360 mg/m2 of doxorubicin or equivalent doxorubicin cardiotoxic dose and/or LVEF (echo or MUGA) < 50%.
6. Known metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, had a negative imaging study within 4 weeks of study entry, is clinically stable with respect to the tumor at the time of study entry, and is not receiving steroid therapy or taper
7. Prior therapy with rapamycin, mTOR inhibitors or tacrolimus
8. Prior anticancer treatment (chemotherapy, radiotherapy, hormonal, immunotherapy, biological response modifiers, signal transduction inhibitors, etc) within 4 weeks prior to the first dose of RAD001; the interval is ≥ 2 weeks for signal transduction inhibitors with a half-life known to be <24 hours, and is ≥ 6 weeks for nitrosourea or mitomycin. The following exceptions are allowed:

   * hormonal therapy (e.g., Megace) for appetite stimulation
   * nasal, ophthalmic, and topical glucocorticoid preparations
   * a stable dose of corticosteroids for at least two weeks
   * low dose maintenance steroid therapy for other conditions
   * physiologic hormone replacement therapy (e.g., thyroid supplementation for thyroid deficiency or oral replacement glucocorticoid therapy for adrenal insufficiency)
9. Pre-existing malabsorption syndrome, irritable bowel syndrome or other clinical situation which could affect oral absorption
10. Ongoing toxicity associated with prior anticancer therapy (except peripheral neuropathy of ≤ grade 1 by NCI toxicity criteria and alopecia)
11. Another primary malignancy within the past three years (except for non-melanoma skin cancer and cervical carcinoma in situ)
12. Known Grade 3 or 4 hypersensitivity to macrolide antibiotics (e.g., clarithromycin, erythromycin, azithromycin)
13. Significant uncontrolled cardiovascular disease
14. Active infection requiring systemic therapy
15. Known HIV infection
16. Inadequate recovery from any prior surgical procedure or having undergone any major surgical procedure within 2 weeks prior to the first dose of RAD001. Patients having undergone recent placement of a central venous access port will be considered eligible if they have recovered
17. Presence of any other life-threatening illness or organ system dysfunction which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluating the safety of the study drug

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-10; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Dose (RD) | 4 weeks
  The Maximum Tolerated Dose (MTD) is defined as the dose in which 2 of 3 or 2 of 6 patients experience a Dose Limiting Toxicity (DLT).The Recommended Dose (RD) is defined as one dose level below the MTD.

SECONDARY OUTCOMES:
Safety profile of drug combination | from the first dose of investigational medication to 30 days after trial end.
  Safety will be assessed by physical examination, interim history, and laboratory assessments. Adverse events will be graded according to the NCI-CTCAE, version 3.0.
Response Rate | every 8 weeks
  For patients with measurable disease overall tumor response is performed according to RECIST criteria. For patients with non measurable disease (prostate and ovarian cancer) response can be assessed according to serum tumor markers (Rustin criteria for CA 125 and criteria for PSA response).
PK parameters | until 14 days post infusion
  PK parameters: terminal half life (T1/2), Total Body Clearance (ClTB), apparent volume of distribution (Vss), Cmax, Tmax, AUC0-48h, AUC0-inf

CONTACTS AND LOCATIONS:
Overall Officials: Cristiana Sessa, MD, Study Chair — Istituto Oncologico della Svizzera Italiana- Ospedale s.Giovanni - 6500 Bellinzona, Switzerland
Locations (3):
- Italy (2):
  - Fondazione IRCSS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
- Istituto Oncologico della Svizzera Italiana, Bellinzona, Switzerland

REFERENCES:
- [Background] Guba M, von Breitenbuch P, Steinbauer M, Koehl G, Flegel S, Hornung M, Bruns CJ, Zuelke C, Farkas S, Anthuber M, Jauch KW, Geissler EK. Rapamycin inhibits primary and metastatic tumor growth by antiangiogenesis: involvement of vascular endothelial growth factor. Nat Med. 2002 Feb;8(2):128-35. doi: 10.1038/nm0202-128. PMID 11821896
- [Background] Pollock Rea: Cell shrinkage, cell cycle arrest and anti-angiogenesis underlie the anti-tumor activity of the m-TOR inhibitor AP23573, AACR-NCI-EORTC International Conference, 2003, pp Abstr. B160
- [Background] Tan C, Cruet-Hennequart S, Troussard A, Fazli L, Costello P, Sutton K, Wheeler J, Gleave M, Sanghera J, Dedhar S. Regulation of tumor angiogenesis by integrin-linked kinase (ILK). Cancer Cell. 2004 Jan;5(1):79-90. doi: 10.1016/s1535-6108(03)00281-2. PMID 14749128
- [Background] Brown NS, Bicknell R. Thymidine phosphorylase, 2-deoxy-D-ribose and angiogenesis. Biochem J. 1998 Aug 15;334 ( Pt 1)(Pt 1):1-8. doi: 10.1042/bj3340001. PMID 9693094
- [Background] Parmar MK, Ledermann JA, Colombo N, du Bois A, Delaloye JF, Kristensen GB, Wheeler S, Swart AM, Qian W, Torri V, Floriani I, Jayson G, Lamont A, Trope C; ICON and AGO Collaborators. Paclitaxel plus platinum-based chemotherapy versus conventional platinum-based chemotherapy in women with relapsed ovarian cancer: the ICON4/AGO-OVAR-2.2 trial. Lancet. 2003 Jun 21;361(9375):2099-106. doi: 10.1016/s0140-6736(03)13718-x. PMID 12826431
- [Background] Stewart, C. F. and Ratain, M. J. Topoisomerase interactive agents. In: V. T. DeVita, Jr., S. Hellman, and S. A. Rosenberg (eds.), Cancer: Principles and practice of oncology, pp. 452-467. Philadelphia: Lippincott-Raven Publishers, 1997.
- [Background] Riggs, C. E. J. Antitumor antibiotics and related compounds. In: M. C. Perry (ed.) The chemotherapy source book, 2nd edition, pp. 345-386. Baltimore: Williams and Wilkins, 1997.
- [Background] Lyass O, Uziely B, Ben-Yosef R, Tzemach D, Heshing NI, Lotem M, Brufman G, Gabizon A. Correlation of toxicity with pharmacokinetics of pegylated liposomal doxorubicin (Doxil) in metastatic breast carcinoma. Cancer. 2000 Sep 1;89(5):1037-47. doi: 10.1002/1097-0142(20000901)89:53.0.co;2-z. PMID 10964334
- [Background] Ranson MR, Carmichael J, O'Byrne K, Stewart S, Smith D, Howell A. Treatment of advanced breast cancer with sterically stabilized liposomal doxorubicin: results of a multicenter phase II trial. J Clin Oncol. 1997 Oct;15(10):3185-91. doi: 10.1200/JCO.1997.15.10.3185. PMID 9336354